CLINICAL TRIAL: NCT06893484
Title: Assessing Completion of Medication Abortion for Very Early Pregnancies
Brief Title: Assessment of Early Pregnancy MAB Completion
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lyndsey Benson, Assistant Professor, Obstetrics & Gynecology, University of Washington
Other Study IDs: STUDY00022025
Record Dates: First submitted 2025-03-09; First posted 2025-03-25 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy; Abortion Early
Keywords: very early pregnancy; pregnancy test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Early Pregnancy: Participants with early pregnancy ≤ 42 days by last menstrual period or ultrasound undergoing a medication abortion will be enrolled.
  Interventions: Diagnostic Test: Weekly high-sensitivity urine pregnancy tests

INTERVENTIONS:
Diagnostic Test: Weekly high-sensitivity urine pregnancy tests — Participants will take a high-sensitivity urine pregnancy test at home weekly for up to 4 weeks compared to the taking just one home urine pregnancy test at 4-5 weeks. Participants will also complete short weekly questionnaires on their pregnancy symptoms and follow-up care.

SUMMARY:
This is a prospective study to evaluate if successful completion of a medication abortion in patients with very early pregnancy can be detected with a urine pregnancy test at 2 weeks instead of 4 weeks. Additionally, the resolution of pregnancy symptoms in these patients will be characterized. Enrolled participants will take take weekly pregnancy tests and complete weekly questionnaires on their pregnancy symptoms for 4 weeks after their medication abortion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant person with early pregnancy ≤42 days
* Eligible and consented to a medication abortion
* Have access to receiving text messages and the internet
* Able to read and understand English

Exclusion Criteria:

- Privacy or safety concerns about filling out the surveys

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll patients who meet the inclusion criteria at clinical sites in Washington, Georgia, and Maryland.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with negative high-sensitivity urine pregnancy test at 2 weeks | From time of taking Mifepristone to negative pregnancy test or 4-5 weeks of questionnaires
  To estimate the proportion of negative high-sensitivity urine pregnancy tests in participants with very early pregnancy and a complete abortion at 2 weeks after taking Mifepristone and compare this proportion to the proportion of negative high-sensitivity urine pregnancy tests in participants with very early pregnancy and a complete abortion at 4 weeks

SECONDARY OUTCOMES:
Time to resolution of pregnancy symptoms | From time of taking Mifepristone to negative pregnancy test or 4-5 weeks of questionnaires
  To compare the timing of pregnancy symptom resolution per patient report on weekly questionnaires with the timing of a negative high-sensitivity urine pregnancy test result

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsey Benson, MD, MS, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Carafem, Atlanta, Georgia
  - Carafem, Chevy Chase, Maryland
  - Cedar River Clinics, Renton, Washington

IPD SHARING:
Plan to Share IPD: No
Access to study IPD will not be shared for this study due to the sensitive, private nature of the clinical care received by participants. Participant safety and confidentiality is of utmost importance for this study.